CLINICAL TRIAL: NCT05723211
Title: The Effects of a 4-week Vinyasa Yoga Program on Sleep and Cardiovascular Health in Adults With Insomnia Symptoms: A Randomized Controlled Trial
Brief Title: The Yoga and Insomnia Study
Acronym: YOGi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Caitlin Cheruka, Graduate Student Researcher, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY22110168
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Insomnia; Insomnia, Psychophysiological; Sleep Disorder
Keywords: sleep; cardiovascular; insomnia; yoga; physical activity
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The research staff conducting the outcome assessments will be blinded to the participant intervention group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vinyasa yoga group (Experimental): The vinyasa yoga practice will be 60 minutes in duration and includes standing, seated, and supine postures in the following sequences in order: integration, sun salutations, crescent lunge series, balancing, standing, back bending, and restorative series. Participants will be instructed to follow the cues provided in the video and to take any necessary modifications to make each yoga pose more accessible. Vinyasa yoga intervention level 1 will be performed for week 1, level 2 will be performed for week 2, and level 3 will be performed for weeks 3 and 4 of the intervention.
  Interventions: Behavioral: Vinyasa yoga group
- Non-active control group (Other): The participants in the non-active control condition will serve as a control group. They will be asked to maintain their current lifestyle habits and refrain from starting a new exercise and/or yoga program. A staff member will contact each participant weekly to check in and review any changes to their medical history or activity levels.
  Interventions: Other: Non-active control group

INTERVENTIONS:
Behavioral: Vinyasa yoga group — Participants will be instructed to perform a pre-recorded 60-minute vinyasa yoga session 3 times a week for 4 weeks.
  Arms: Vinyasa yoga group
Other: Non-active control group — Participants will be instructed to sit quietly for 60 minutes and watch a nature documentary during this time. The participants will be asked to maintain their current lifestyle habits and refrain from starting a new exercise and/or yoga program.
  Arms: Non-active control group

SUMMARY:
The purpose of our study is to examine the effects of a 4-week vinyasa yoga program on sleep-related and cardiovascular outcomes in adults with insomnia symptoms. This study will examine the following aims:

To examine the effects of a 4-week vinyasa yoga program compared to a non-active control condition on subjective and objective sleep-related outcomes in adults who report insomnia symptoms.

To examine the effects of a 4-week vinyasa yoga program compared to a non-active control on cardiovascular health.

To examine the effects of a single session of vinyasa yoga compared to a non-active control condition on sleep- and cardiovascular-related outcomes collected overnight.

Researchers will compare the yoga group and the non-active control group to see if there are any improvements in sleep and cardiovascular health.

DETAILED DESCRIPTION:
This study will examine the effects of a 4-week vinyasa yoga program on sleep-related and cardiovascular outcomes using a randomized parallel group design. Following baseline assessments, participants will be randomly assigned into one of the two experimental conditions (i.e., vinyasa yoga, non-active control condition) based on stratification by sex (i.e., male, female) in a 1:1 ratio.

All groups will complete an initial in-person experimental session during the early evening: those in the vinyasa yoga group will be guided through a supervised vinyasa yoga session and those in the non-active control group will complete a quiet rest session. Participants will be provided an Actiwatch and heart rate monitor to measure acute experimental effects on sleep and nocturnal heart rate variability.

Following the initial supervised session, those in the vinyasa yoga intervention will be provided with a yoga mat and a standardized video and asked to practice 3 times per week for 4 weeks; compliance will be monitored by an online log. The non-active control group will not receive any yoga intervention and will be asked to avoid starting a new exercise routine.

Following the 4-week intervention, all participants will complete post-intervention sleep and cardiovascular assessments following the same procedures used at baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Insomnia Severity Index (ISI) score ≥ 10
2. Age 18-55 years
3. Insufficiently active defined by the Stanford Leisure-Time Activity Categorical Item responses below public health physical activity guidelines

Exclusion Criteria:

1. Self-reported regular vinyasa and/or power yoga practice defined as ≥ 60 minutes/week within the past 3 months
2. Diagnosed medical condition requiring medical clearance defined as a 'yes' response on follow-up questions pertaining to a present medical condition(s) via Physical Activity Readiness Questionnaire for Everyone (PAR-Q+)
3. Physical limitations and/or mobility restriction that would interfere with the ability to perform yoga defined as a 'yes' response on the PAR-Q+; self-reported lack of treatment for a major psychiatric disorder via medical history survey
4. High risk for obstructive sleep apnea defined as score ≥ 5 via STOP-Bang score
5. Self-reported current pregnancy or planning to become pregnant within the next 3 months
6. Overnight shift work defined as regularly working any time between 00:00 and 06:00 am
7. Self-reported current treatment for insomnia via medical history survey
8. Medications that may affect heart rate during exercise via self-report on the medical history survey

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index | Baseline, post-intervention (4 weeks)
  Insomnia Severity Index is a 7-item self-report questionnaire that assesses the severity of the nighttime and daytime impact of insomnia symptoms. Each question is rated on a 5-point Likert scale, with a score of 0 indicating 'no problem' and 4 indicating 'very severe'. The total score is obtained by summing the scores of the individual items ranging from 0 to 28; a higher score indicates more severe insomnia symptoms.
Change in nocturnal root mean square of successive difference between normal heartbeats (RMSSD) | Baseline, post-intervention (4 weeks)
  Nocturnal root mean square of successive difference between normal heartbeats will be assessed for 1 night with a Polar heart rate monitor strap; an increase indicates better cardiovascular health

SECONDARY OUTCOMES:
Change from baseline sleep efficiency at 4 weeks | Baseline, post-intervention (4 weeks)
  Actigraphy-assessed sleep efficiency, averaged over 7 nights
Change from baseline total sleep time at 4 weeks | Baseline, post-intervention (4 weeks)
  Actigraphy-assessed total sleep time, averaged over 7 nights
Change from baseline resting systolic blood pressure at 4 weeks | Baseline, post-intervention (4 weeks)
  Resting systolic blood pressure will be measured using an automated blood pressure system in the seated position
Change from baseline resting heart rate at 4 weeks | Baseline, post-intervention (4 weeks)
  Resting heart rate will be measured using a automated blood pressure system in the seated position
Change from baseline resting carotid-femoral pulse wave velocity | Baseline, post-intervention (4 weeks)
  Pulse wave velocity is a measure of arterial stiffness
Change from baseline quality of sleep | Baseline, post-intervention (4 weeks)
  Sleep quality will be assessed using a sleep diary on a scale of 'very poor' to 'very good'
Change from baseline in Epworth Sleepiness Scale | Baseline, post-intervention (4 weeks)
  Daytime sleepiness will be measured using the Epworth Sleepiness Scale (ESS). It is a brief 8-item questionnaire asking individuals to rate the likelihood of falling asleep on a 4-point scale (0 indicating 'would never doze off' and '3' indicating 'high chance of dozing') across eight situations that occur in daily life. The scores are summed for a total score that ranges from 0-24; a score ≥ 10 indicating clinically significant daytime sleepiness.
Change from baseline in Ford Insomnia Response to Stress Test | Baseline, post-intervention (4 weeks)
  Sleep reactivity, the stress-related vulnerability to experience sleep disturbances under stressful conditions will be measured by the Ford Insomnia Response to Stress Test; higher scores are associated with more sleep difficulties and elevated physiological stress.
Change from baseline in Patient Health Questionnaire | Baseline, post-intervention ( 4 weeks)
  Depression severity will be measured using the Patient Health Questionnaire which assess depressive symptoms over the past two weeks; a score > 10 indicates moderate severity depression symptoms.
Change from baseline in Generalized Anxiety Disorder-7 Questionnaire | Baseline, post-intervention (4 weeks)
  Anxiety severity will be measured using the Generalized Anxiety Disorder Questionnaire which assess symptoms over the past two weeks; a score ≥ 10 detects generalized anxiety disorder.

OTHER OUTCOMES:
Sleep efficiency | Immediately after first intervention session (1 night)
  Mean actigraphy-assessed sleep efficiency will be immediately assessed after the initial session of the intervention for 1 night
Total sleep time | Immediately after first intervention session (1 night)
  Mean actigraphy-assessed total sleep time will be immediately assessed after the initial session of the intervention
Nocturnal root mean square of successive difference between normal heartbeats | Immediately after first intervention session (1 night)
  Nocturnal root mean square of successive difference between normal heartbeats will be assessed immediately after the first intervention session for 1 night; an increase value indicates better cardiovascular health
Change in acute anxiety symptoms | pre- and post-initial intervention session
  Acute anxiety symptoms will be measured using the State-Trait Inventory 20-item pre- and post-initial first intervention session
Change in mood | pre- and post-initial intervention session
  Acute changes in mood will be measured using the Profile of Mood States brief form. This will assess the feelings of tension, depressed mood, energy, fatigue, and total mood disturbances based on how the participant feels right now using a 5-point Likert scale ranging from 0 "not at all" to 4 "extremely
Change in percent body composition | baseline, post-intervention (4 weeks)
  Body composition will be measured using the bio-electrical impedance; a decrease in percentage indicates improved body composition

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin A. Cheruka, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual deidentified data that are relevant to the primary aims of the study will be provided by external researchers along with a relevant data dictionary.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 1 year following peer-reviewed publication of research questions outlined in the specific aims and ending 5 years following publication of study results
Access Criteria: Data access will be provided to external researchers who provide a methodologically sound proposal for secondary data analysis that is approved by the investigators of the study. Proposals should be directed to the study PI.